CLINICAL TRIAL: NCT06173440
Title: Management of an Imipenem-resistant Acinetobacter Baumannii Alert in a French University Hospital: A Retrospective Study
Brief Title: Management of an Imipenem-resistant Acinetobacter Baumannii Alert in a French University Hospital
Acronym: Baumannii
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7588
Record Dates: First submitted 2022-11-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Acinetobacter Baumannii
Keywords: Acinetobacter baumannii; Imipenem-resistant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colonization with imipenem-resistant Acinetobacter baumannii (IBA) is an unfavorable event for the patient, especially in intensive care. Indeed, it exposes the patient to the risk of developing serious infections, extremely difficult to treat. ABRI is a particularly resistant bacterium in the environment. When an ABRI epidemic occurs in a department as central to the hospital as a surgical resuscitation department, the control of such an event can be extremely complex. There are few clear and detailed descriptions in the literature of how to manage this type of outbreak, let alone an ABRI outbreak of this magnitude.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Patient having been hospitalized in the surgical resuscitation service of Hautepierre during the ABRI epidemic, between 01/05/2015 and 01/01/2019 inclusive and having been colonized and/or infected by ABRI (according to bacteriological results transmitted to the hygiene service).
* Subject having given his/her agreement, after information, for the reuse of his/her data for the purpose of this research

Exclusion criteria:

* Subject having expressed his opposition to participate in the study
* Subject under guardianship or curatorship
* Subject under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) having been hospitalized in the surgical resuscitation service of Hautepierre during the ABRI epidemic, between 01/05/2015 and 01/01/2019 inclusive and having been colonized and/or infected by ABRI
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the management of an imipenem-resistant Acinetobacter baumannii outbreak that occurred from 2015 to 2019 in a surgical intensive care unit | Through study completion, an average of 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service Equipe opérationnelle d'hygiène - CHU de Strasbourg - France, Strasbourg, France